CLINICAL TRIAL: NCT01016093
Title: Zoledronic Acid for the Prevention of Bone Loss Post-bone Marrow Transplantation for Thalassemia Major Patients: A Prospective Pilot Study
Brief Title: Zoledronic Acid for the Prevention of Bone Loss Post-bone Marrow Transplantation for Thalassemia Major Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: Novartis (Industry)
Responsible Party: Mahdi Jalili MD / Hematology-Oncology and SCT Research Center, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HORCSCT-0601
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Beta-Thalassemia; Bone Marrow Transplantation
Keywords: Thalassemia; BMT; HSCT
MeSH Terms: conditions — beta-Thalassemia; Thalassemia | interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Patients in this arm received zoledronic acid.
  Interventions: Drug: Zoledronic acid
- Control (Placebo Comparator): Patients in this arm received placebo as control group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zoledronic acid — Zoledronic acid 4 mg adjusted dose based on renal function IV 15-minute infusion every 3 months for a total of one year ( 4 doses ) beginning as soon as possible after randomization.
  Other Names: Zometa
  Arms: Intervention
Drug: Placebo — Placebo
  Arms: Control

SUMMARY:
This is prospective randomized, double blind study designed to evaluate the use of zoledronic acid in the prevention prevention of bone loss post allogenic BMT done for beta-thalassemia major patients.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* Patients must be 18 years old and over.
* Diagnosed with beta-thalassemia major
* Scheduled for allogenic bone marrow transplantation
* The date of randomization must be no more than 1 week after BMT.
* Patients must be accessible for follow-up.
* Life expectancy of at least 12 months from randomization.

Exclusion Criteria:

* Patients with any clinical or radiological evidence of existing fracture in the lumbar spine and/or total hip.
* Patients with a history of fracture with low-density or no associated trauma.
* Osteoporotic patients with T-score <= -2.5
* Previous treatment with a bisphosphonate.
* Patients with abnormal renal function as evidenced by either a serum creatinine determination 1.5 x or greater above the upper limit of normal or by a calculated creatinine clearance of 30 ml/minute or less.
* Pregnancy and lactation.
* Women of childbearing potential not on a medically recognized form of contraception.
* Subjects who, in the opinion of the investigator, are unlikely to cooperate fully during the study.
* Subjects participating simultaneously in studies with unapproved drugs, indications or treatment regimens.
* Known hypersensitivity to zoledronic acid or bisphosphonates.
* Patients with prior exposure to anabolic steroids, growth hormone, Parathyroid Hormone (PTH) or other drugs known to affect the skeleton (e.g., calcitonin, mithramycin, or gallium nitrate).
* Serious intercurrent illness
* History of metabolic bone diseases
* History of corticosteroid treatment for other causes
* History of antiepileptic drug treatment
* History or surgery at the lumbosacral spine, with or without implantable devices.
* Any disease of the spine that would preclude the proper acquisition of a lumbar spine DXA.
* Mental illness that precludes the patient from giving informed consent.
* Current active dental problems including infection of the teeth or jawbone (maxilla or mandibular); dental or fixture trauma, or a current or prior diagnosis of osteonecrosis of the jaw (ONJ), of exposed bone in the mouth, or of slow healing after dental procedures.
* Recent (within 6 weeks) or planned dental or jaw surgery (e.g.. extraction, implants)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-11 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
To describe the percent change in the lumbar spine (L1 to L4) BMD, as measured by dual energy X-ray absorptiometry, at 12 months in patients with beta-thalassemia major undergoing allogenic BMT randomized to zoledronic acid versus placebo. | 1 year

SECONDARY OUTCOMES:
To describe the percent change in total hip BMD at 12 months in the two study arms. | 1 year
To compare the changes in bone turn over markers at 3, 6, and 12 months in the two treatment arms. | 1 year
To describe the incidence rate of all clinical fractures at 1 year in the two study arms. | 1 year
To describe the general safety of zoledronic acid. | 1 year
To describe the percent change in lumbar spine (L1 to L4) BMD and total hip BMD at 6 months when available. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Hematology-Oncology & SCT Research Center, Tehran, Tehran Province, Iran